CLINICAL TRIAL: NCT03929614
Title: Development and Validation of the MOBI Questionnaire
Acronym: MOBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Hubert Labelle, MD, Orthopedist and Principal Investigator, St. Justine's Hospital
Other Study IDs: 2018-1756
Record Dates: First submitted 2019-04-02; First posted 2019-04-29 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Idiopathic Scoliosis
Keywords: Brace Treatment; Health-related quality of life (HRQOL); Questionnaire development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MOBI validation — Final version will be distributed to 176 French speaking subjects, 30 of whom are randomly selected and will fill it a second time, at after 72 hrs. To consider of its kind, Moreover, the Bem Inventory for Children will be completed by everyone as well as the SF-12 and SRS-22.

SUMMARY:
Scoliosis is a common spinal deformity in adolescents. Orthopedic brace treatment is the only conservative (nonsurgical) treatment effective in limiting the progression of this deformity. It is a difficult treatment for young people (discomfort, self-image, limitation in activities) who must wear this rigid orthosis between 20-23 hrs / day during the growth spurt. Recent studies have shown that the effectiveness of this treatment is related to the wearing time of the corset. However, there is a serious problem of compliance to treatment. On average, the brace is worn only 12 hrs / day. A negative perception of the patient with respect to the brace can lead to treatment failure if the brace is not worn. It is therefore essential to understand the impact of the brace on the quality of psychological life, the daily activities and the comfort of young patients. Unfortunately, there is no valid instrument to evaluate all these dimensions. The objective of this project is to develop a questionnaire that can measure the quality of life of patients wearing a brace and validate it for its clinical use.

The investigators have created a questionnaire based on the best knowledge published on the subject, opinions of experts in the field and a group of patient partners.

At the end of this project, a questionnaire will be available for the first time to assess in depth the perception that patients have of their braces. It can be used to adjust braces in the clinic, as well as to support and encourage compliance to the treatment

DETAILED DESCRIPTION:
Increase treatment adherence by 50%: 1- by identifying the reasons of non-adherence with MOBI, the first bilingual quality of life (QL) measurement questionnaire dedicated to braces, 2- using for the first time a Multidisciplinary Support Team (MST) for the patient / family.

The BrAIST study showed an inverse correlation between the duration of brace wear and the probability of progression, a wearing time of 0 to 6 hrs / day with a proportion at 59% progression ≥50 ° vs 7% for a brace wear> 17 hours. Knowing that the average daily brace wear duration measured is much lower than that prescribed, there is a problem of compliance whose in which the causes are unknown. Unsuitable questionnaires assessed the QoL of AIS patients on TLSO and have reflected the impact of the disease on psychological health, perceptions of self-image and daily activities, but do not isolate the factors associated with non-compliance to TLSO. In addition, there is no biopsychosocial intervention strategy in care settings to improve compliance.

The investigators have expertise in this field since the investigator have carried out cross-cultural adaptation and validation of 2 QL instruments in the AIS. In addition, the investigator and his team developed a body diagram to evaluate the comfort of patients under brace treatment and correlated with pressure measurements at the skin-brace interface. The investigator's also used in a previous RCT thermal sensors to measure the wearing time of the braces.

The investigator's team propose to develop and validate MOBI (My Orthopedic Brace Inventory), the first bilingual multidimensional QL questionnaire dedicated to the wearing of the brace to measure the physical and functional well-being, emotional and social wellness. We will use MOBI to identify the elements associated with non-compliance to TLSO and for the first time in the world MST, a multi-disciplinary team (nurse, orthotist, psychologist, social worker) to intervene on the 4 identified dimensions, with the assumption that this intervention will improve by 50% the wearing time of the brace.

ELIGIBILITY:
Inclusion Criteria:

* AIS.
* 10-16 years old, with brace treatment.
* Ability to read and understand English or French.
* Physical and mental ability to adhere to bracing protocol.

Exclusion Criteria:

* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature.
* Patients with symptom of a neurological disorder.
* Patients with any other disorder of the musculoskeletal system affecting the lower limbs,

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: AIS patients with brace treatment.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Score distribution for the new MOBI questionnaire scales | At baseline (at recruitment)
  To develop a self-report questionnaire to assess the quality of life of scoliotic children treated by a Boston brace. There are 6 sub scales : Emotional well-being (7 items, sub score between 0 and 28, best score is 0); Functional well-being (6 items, subscore between 0 and 24, best score is 0); Physical well-being (4 items, subscore between 0 and 16, best score is 0); Social well-being (6 items, subscore between 0 and 24, best score is 0); Barriers related to Patient (4 items, subscore between 0 and 16, best score is 0); Barriers related to System (3 items, subscore between 0 and 12, best score is 0); Barriers related to Treatment (3 items, subscore between 0 and 12, best score is 0). Total score of the MOBI score is obtained by summing the subscores of all subscales (between 0 and 136, best score is 0).
Internal validity, scale MOBI | At baseline (at recruitment)
  Chronbach's alpha coefficient, measured at the first visit and at the second visit.
The test-retest reliability of MOBI questionnaire | At baseline (at recruitment)
  The test-retest reliability of MOBI will be evaluated using the intraclass correlation coefficient with about 72 hours interval.
The structural validity of the MOBI questionnaire | At project completion (up to 48 months upon recruitment)
  Principal component analysis with factor extraction to identify the factorial structure of the MOBI questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Labelle, MD, Principal Investigator — Ste Justine's
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided